CLINICAL TRIAL: NCT04196049
Title: Removal of Massive Subretinal Organized Blood Clot With Fragmatome
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, medical doctor, Changhua Christian Hospital
Other Study IDs: 191203
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Age-Related Macular Degeneration
Keywords: organized blood clot; fragmatome; exudative age related macular denegeration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: fragmatome — Patients with massive subretinal hemorrhage from age related macular degeneration and organized subretinal blood clot were managed by inferior retinectomy. The subretinal organized blood clot was dragged to the preretinal space and removed by fragmatome. The retinal was reattached with perfluorocarbon liquid and laser was applied at the margin of retinectomy. Silicon oil was infused at the end of surgery.

SUMMARY:
By using the ultrasound power delivered by fragmatome, the hard, organized blood clot could be removed easily.

ELIGIBILITY:
Inclusion Criteria:

* Patients with massive subretinal hemorrhage from age related macular degeneration
* Patients had organized subretinal blood clot were managed by inferior retinectomy.

Exclusion Criteria:

* Patients without massive subretinal hemorrhage
* Patients were not age related macular degeneration.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with massive subretinal hemorrhage from age related macular degeneration and organized subretinal blood clot were managed by inferior retinectomy
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Visual acuity | Before operation, 1 weeks after operation, 1 month after operation.
  visual acuity change in logMAR in different time point
spherical equivalent | Before operation
  spherical power + half of cylinder power

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan